CLINICAL TRIAL: NCT00299884
Title: The Comparison of the Efficacy of Ezetimibe and Fenofibrate Versus Atorvastatin Alone in the Lowering of LDL Cholesterol
Brief Title: Atorvastatin Versus Ezetimibe and Fenofibrate as a Lipid-lowering Strategy
Status: Completed | Type: Observational
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Stephen LaHaye, Principal Investigator, Queen's University
Other Study IDs: DMED-816-04
Record Dates: First submitted 2005-09-09; First posted 2006-03-07 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Dyslipidemia; Vascular Disease
Keywords: Randomized; non-blinded; prospective; open-label; LDL-C; HDL-C
MeSH Terms: conditions — Dyslipidemias; Vascular Diseases | interventions — Atorvastatin; Fenofibrate

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Apo-lipo B
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Lipitor 20 mg
  Interventions: Drug: Lipitor 20 mg
- 2: Lipidil Supra 160 mg and Ezetrol 10 mg
  Interventions: Drug: Combination Ezetrol 10 mg and Lipidil Supra 160 mg

INTERVENTIONS:
Drug: Lipitor 20 mg — A/A for 6 weeks
  Groups: 1
Drug: Combination Ezetrol 10 mg and Lipidil Supra 160 mg — a/a for 6 weeks
  Groups: 2

SUMMARY:
The primary aim of this study is to evaluate the efficacy and non-inferiority of a lipid-lowering medication regimen comprised of the medications ezetimibe and fenofibrate taken daily, versus atorvastatin daily in lowering levels of low-density lipoprotein (LDL-C) cholesterol. Additionally, other aims would include effects on other types of blood cholesterol and examining the safety of the ezetimibe and fenofibrate regimen, as compared to atorvastatin.

DETAILED DESCRIPTION:
It has been demonstrated in several previous primary and secondary studies that lowering low-density lipoprotein cholesterol (LDL-C) with the use of medications such as 3-hydroxy-3-methylglutaryl-coenzyme A (HMG-CoA) reductase inhibitors improves mortality and morbidity related to cardiovascular events in patients with hypercholesterolemia. Such inhibitors, which are known as 'statins', act to block the synthesis of cholesterol in the liver. These medications are generally well tolerated by the vast majority of patients, but a small number experience side effects, most seriously those of myopathies, rhabdomyolysis and elevated liver enzymes - recognition of this fact, that statins are not universally without problems, highlights the need for viable alternatives.

Ezetimibe is a relatively new medication in Canada, approved for use in patients with cholesterol problems. It is an intestinal cholesterol binder that is known to be well-tolerated, with side effects similar to placebo. Alone, it has a modest effect in the lowering of LDL-C. Fenofibrate is a medication that also works through the liver and has long been used to adjust blood lipid levels in patients with mixed lipid problems. Alone it also has a modest effect in the lowering of LDL-C. Recent study, however, has shown that the effect of ezetimibe and fenofibrate together in the lowering of LDL-C is greater than that of either drug alone. This combination, if as effective in this regard as atorvastatin, would prove a valid alternative to the use of the atorvastatin in the lowering of LDL-C, and a benefit for patients who have had problems tolerating statin therapy but still require medication for elevated cholesterol.

ELIGIBILITY:
Inclusion Criteria:

-Study is confined to subjects with elevated LDL-C levels 3.0 mmol/L and greater.

Exclusion Criteria:

* Abnormal liver enzymes (ie, AST, ALT greater than three times the upper limit of normal);
* Creatine kinase levels more than two times the upper limit of normal;
* Uncontrolled ethanol use (this may affect compliance);
* Pregnant or breastfeeding women or women not using adequate contraceptive methods;
* Previous history of intolerance or adverse effects with statins;
* Previous history of intolerance or adverse effects with fibric acid derivatives;
* Previous history of intolerance or adverse effects with ezetimibe;
* Uncontrolled diabetes (HbA1c > 10%);
* Recent myocardial infarction (within 6 weeks);
* Concurrent enrollment in another study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects aged 18-85 with elevated LDL-C levels 3.0 mmol/L and greater.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2005-01; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
To examine the efficacy of a combination of ezetimibe and fenofibrate in comparison with that of atorvastatin in lowering LDL-C. | 12 weeks

SECONDARY OUTCOMES:
To examine the efficacy of a combination of ezetimibe and fenofibrate in comparison with that of atorvastatin in lowering triglyceride levels, raising HDL-C levels and lowering of hsCRP levels. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A LaHaye, MD, Principal Investigator — Vascular Disease Prevention and Research Centre
Locations (1):
- Vascular Disease Prevention and Research Centre, Hotel Dieu Hospital, Kingston, Ontario, Canada